CLINICAL TRIAL: NCT05837559
Title: Randomized Study of the Traditional WHO Partograph and Korle-Bu Modified WHO Partograph for Uncomplicated Labour
Brief Title: Traditional WHO Partograph and Korle-Bu Modified WHO Partograph for Uncomplicated Labour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ghana Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHS-ET/M.2-P5.2/2020-2021
Record Dates: First submitted 2023-01-26; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-02

CONDITIONS: Labor Complication
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional WHO Partograph for Uncomplicated Labour (Active Comparator): With the Traditional WHO partograph, uterine contractions will be assessed every 30 minutes, fetal heart will be assessed every 30 minutes and maternal pulse 30 minutes, blood pressure is recorded every 4 hourly and temperature is recorded every 2 hourly. Urine output is recorded every time urine is passed. The woman is encouraged to pass urine every 2 hourly in labour and each specimen is tested for protein and ketones. Drugs, IV fluids, Drugs (Oxytocin) are recorded in the space provided.
  Interventions: Other: Korle-Bu Modified WHO Partograph for Uncomplicated Labour
- Korle-Bu Modified WHO Partograph for Uncomplicated Labour (Experimental): With the Korle-Bu modified partograph, uterine contractions will be assessed every hour (60 minutes), fetal heart will be assessed every 30 minutes and maternal pulse every hour. All other assessments remain as for the traditional partograph.
  Interventions: Other: Korle-Bu Modified WHO Partograph for Uncomplicated Labour

INTERVENTIONS:
Other: Korle-Bu Modified WHO Partograph for Uncomplicated Labour — Monitoring of labour using the Korle-Bu Modified WHO Partograph for Uncomplicated Labour

SUMMARY:
Brief Background:

The partograph is a graphical representation of the events in the first stage of labour. It is an instrument used in monitoring the well being of both the pregnant woman and her fetus (es) as they go through the first stage of labour.

Most studies found the completion of a partograph in a client's record as the exception rather than the norm. Even at urban maternity wards as low as 5% completion rates of partograph have been recorded and in more than 60% of deliveries the partographs were completed after the deliveries, indicating it was being utilized only as a record-keeping procedure, not as a monitoring tool. The correct and effective use of the partograph is in itself labour intensive even with the requisite skills, making it unfriendly to use in situations where the delivery rates are high with few skilled attendants

General Aim:

To determine whether the use of a Korle-Bu modified WHO partograph will result in similar or improved patronization and leading to consistent monitoring of first stage labour and better outcomes compared to the traditional WHO partograph.

Methods: This will be a randomized study of women presenting in labour with uncomplicated pregnancies to the Korle-Bu Teaching and La General hospitals in Accra. 500 labouring women will be monitored with the traditional WHO partograph in one arm and 500 labouring women will be monitored with the Korle-Bu modified WHO partograph. Computer generated cluster randomization with concealment will be used in patient selection and same research assistants ( Residents and Nurses) will be trained to stick to patient specific protocols for labout monitoring. Variables to be collected besides sociodemographic and obstetric data will include duration of labour, any interventions and neonatal and maternal outcome.

Expected outcome (Expected results/what you hope to achieve from the study):

It is expected that the Korlebu Teaching Hospital (KBTH) modified WHO partograph will be more user friendly, making it easier for service providers to use as a labor management tool than the traditional WHO partograph as intended, to reduce perinatal complication.

DETAILED DESCRIPTION:
Background:

The partograph which is a graphical representation of the events in the first stage of labour is a prospective instrument used in monitoring the well being of both the pregnant woman and her fetus (es) as they go through the first stage of labour. Primarily it is to prevent prolonged labour and its attendant adverse outcomes for both mother and baby.

It provides timely information regarding further intervention in the form of referral to a higher-level facility, labour augmentation, and caesarean section etc. depending upon the resources available. At the same time it facilitates ongoing evaluation of the effects of these interventions. It is also a retrospective guide as to how well or not labour may have been managed. World Health Organization designated management of labour with the Partograph as one of the essential elements of obstetric care at the first referral level.

The correct and effective use of the partograph is in itself labour intensive even with the requisite skills, this makes it unfriendly to use in situations where the delivery rates are high with few skilled attendants.

Problem Statement Worldwide the use of the WHO partograph (Pt) has been very limited especially in low resource centres. Studies have found the completion of a partograph in a client's record was the exception rather than the norm. Even at urban maternity wards as low as 5% completion rates of partograph have been recorded and in more than 60% of deliveries the partographs were completed after the deliveries, indicating it was being utilized only as a record-keeping procedure, not as a monitoring tool. The paucity of use and incorrect use of the partograph could be attributed largely to the fact that it is not simple enough, labour intensive and the minimal staffing at low resources areas. This could result in insufficient monitoring leading to perinatal complication.

Justification/Relevance Decreasing the frequency of examinations and measurements to be made on the partograph for uncomplicated pregnancies and labours will make it more user friendly and making it easier for service providers to use as a labor management tool than the WHO partograph as intended, to reduce perinatal complication. . Findings from this study could justify the use or not of the Korle-Bu modified WHO partograph, which is less labour intensive, as a recommended monitoring tool for uncomplicated labour Hypothesis (if any) Null Hypothesis (Ho) The "Korle-Bu modified" WHO partograph would not lead to a lower proportion of prolonged labour and adverse perinatal outcomes compared to the traditional WHO partograph.

H0: Pm > Pt; H1: Pm ≤ Pt General Objective: To determine whether the use of a Korle-Bu modified WHO partograph will result in similar or improved patronization and better first stage labour outcomes compared to the traditional WHO partograph.

Specific objectives are to:

1. Determine provider's preference of the two partographs ( Pt or Pm).
2. Determine the detection rates of labour complications (slow progress, fetal distress),
3. Determine timing of intervention for labor complications
4. Determine perinatal outcomes (Fresh Stillbirths and APGAR Scores among live births)

Study design:

This study will be randomized trial

Variables:

Variables under study will include:

Main outcome variables: Duration of Labour and comparable perinatal results for mothers as well as consistency in usage of partographs for assistants.

Other variables:

Obstetric characteristics: Parity, Previous mode of delivery, gestational age. Labour characteristics: Duration of first stage of labour, augmentation, mode of delivery, APGAR scores, indication for any interventions and any maternal and neonatal complications.

Demographic background variables: Age, level of education, occupation, marital status, religion, height, weight.

Sample size calculation:

Using Epi Info 3.4.3 with the following assumptions;

* 95% CI and a Power of 80%, With a Ratio of 1:1
* Expected freq of prolonged labour with traditional partograph = 5%
* Expected freq of prolonged labour with modified partograph= 10% Minimum Sample size calculated and adjusted by 5% = 498 and rounded up to 500 for each arm.

Sampling method:

Procedure:

Participants shall be recruited into the study using a cluster randomization. With a sample size of 500 a computer generated random clusters of 5 participants per cluster will give100 clusters and within each cluster all participants shall be selected as per the generated random numbers into the arms with concealment. The concealment is to eliminate selection bias by staff into any of the arms.

Patients who report in labour with a cervical dilatation of between 4 cm and 6 cm who have consent to participate in the study prior to active labour ( Less the 4 cm cervical delectation) will be randomized into 2 groups. Group A will be monitored on the traditional or regular partograph ( Pt) and Group B will be monitored on the Korle-Bu modified partograph (Pm) . The same research assistants (residents and midwives ) will be trained to stick to patient specific protocols for labour monitoring. With the Korle-Bu modified partograph, uterine contractions will be assessed every hour (60 minutes), fetal heart will be assessed every 30 minutes and maternal pulse every hour. All other assessments remain as for the traditional partograph.

Data collection techniques and tools:

Data collection techniques:

Quantitative techniques will be employed using interviewer administered structured questionnaire and observations of the recordings on the partograph.

Close-ended questions will be used and questionnaire designed with appropriate modifications based on literature review of similar studies done elsewhere especially other developing countries or within the country

Data collection tools:

Structured questionnaire and filling up the , Korle-Bu modified WHO or Traditional WHO partographs. Labour will be monitored and adverse outcomes would be identified and addressed just as the traditional WHO partograph. The instrument is only a monitoring aid and decision on intervention during labour are individualized and taken by the obstetrician / service provider conducting the labour.

Data quality control:

Data will be carefully checked for completeness and for any inconsistencies for each question. Any incompleteness and or inconsistencies will be sorted out and doubly entered same day as they are collected. This will help ensure accuracy of data. The study results will be monitored quarterly in terms of time and sample size This will be done by the heads of Departments of Obstetrics and Child Health which shall consist of a 4 member team including the heads for review quarterly.

Pretesting of questionnaire:

Pretesting of tools will be done at Mamprobi Polyclinic labour wards and appropriate modifications will be made to address any concerns before final print out of questionnaire.

Training of interviewers (residents or midwives):

Midwives from both centers and some residents from KBTH will be trained in administering the questionnaire and on the use and completion of the two types of partograph. The assistants' performance and consistency in filling the partographs will also be assessed after the study without their prior knowledge.

Data handling:

Data will be stored at a secure place and Pre- coded soft data will be analyzed with SPPS 21 and presented in text, tables and graphs.

Statistical Analysis:

Frequencies and means will be calculated for continuous variables The Chi-square statistic for categorical data and statistical significance will be set at p< 0.05.

Contingency tables and logistic regressions would be used to examine associations

DISSEMINATION OF RESULTS The results from this study will be presented at the Department of Obstetrics and Gynecology, School of Medicine and Dentistry (KBTH), College of Health Science, at local and international conferences and will be submitted for publishing in peer review journals.

ELIGIBILITY:
Inclusion Criteria:

• Women of parity 0-4 with uncomplicated singleton pregnancy admitted at the maternity wards with live fetus in cephalic presentation at term without contraindication to vaginal delivery NB: Uncomplicated pregnancy- absence of chronic medical conditions and obstetric conditions such IUGR, congenital anomalies

Exclusion Criteria:

* Women in advanced labour ( cervical dilation 6 or more)I
* Induced labour

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Duration of first stage of Labour | 8 hours
  Time of active labour to delivery
Perinatal results | one week
  Apgar scores of babies and admission to NICU. Minimum Apgar score equals 1. Maximum Apgar score equals 10. Higher scores mean better outcome
consistency of use of the partograph | Through study completion. An average of one year
  Percentage of partographs that are completely and appropriately filled

CONTACTS AND LOCATIONS:
Overall Officials: Kareem Mumuni, MD,MPH,FWACS, Principal Investigator — University of Ghana Medical School; Ali Samba, MD, FWACS, Principal Investigator — University of Ghana Medical School; Samuel A Oppong, MD, FWACS, Principal Investigator — University of Ghana Medical School; Kwaku Asah-Opoku, MD,MPH,FWACS, Principal Investigator — University of Ghana Medical School; Michael Y Ntumy, MD,FWACS, Principal Investigator — University of Ghana Medical School; Theodor K Boafor, MD, FWACS, Principal Investigator — University of Ghana Medical School; Kwame Adu-Bonsaffoh, MD, FWACS, Principal Investigator — University of Ghana Medical School; Mercy A Nuamah, md,PhD, Principal Investigator — Family Health Medical School
Locations (1):
- Korle-Bu Teaching Hospital, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December, 2023 and for a year
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] 1 Alaudin Md, Runa Bal, Arunangsu De, Parthajit Mandal, M ayoukh Chakraborty. Monitoring of labor with WHO modified partgram- A stutdy report. Njog 2008; 3: 8-11
- [Background] 2 Beenu Kushwah, Alok Pratap Singh, Shipra Singh. "The Partograph: an Essential Yet underutilized Tool". Journal of Evolution of Medical and Dental Sciences 2013; Vol2, Issue 24, June 17; Page: 4373-4379.
- [Background] 5 Kitila SB, Gmariam A, Molla A, Nemera G (2014) Utilization of Partograph during Labour and Birth Outcomes at Jimma University. J Preg Child Health 1: 101. doi:10.4172/jpch.1000101
- [Background] 6 Mugerwa, KY and Others (2008) Regional Centre for Quality of Health Care. African Midwives Research Network. East Africa. Kenya.
- [Result] FRIEDMAN E. The graphic analysis of labor. Am J Obstet Gynecol. 1954 Dec;68(6):1568-75. doi: 10.1016/0002-9378(54)90311-7. No abstract available. PMID 13207246
- [Result] Gans-Lartey F, O'Brien BA, Gyekye FO, Schopflocher D. The relationship between the use of the partograph and birth outcomes at Korle-Bu teaching hospital. Midwifery. 2013 May;29(5):461-7. doi: 10.1016/j.midw.2012.03.002. Epub 2012 Nov 9. PMID 23146139